CLINICAL TRIAL: NCT04765644
Title: Arginine Supplementation to Improve Cardiovascular and Endothelial Function After NSAID Treatment (ASCENT)
Brief Title: Arginine Supplementation to Improve Cardiovascular and Endothelial Function After NSAID Treatment
Acronym: ASCENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 18IC4757
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: NSAID; Endothelial function; COX-2; Celecoxib; biomarker
MeSH Terms: interventions — Celecoxib; Arginine

STUDY DESIGN:
Intervention Model Description: Healthy male volunteers will be blinded and randomized to 7 days' treatment with celecoxib (200mg bd) or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Celecoxib (Active Comparator): Phase 1: Twenty volunteers will receive celecoxib 200 mg, 2 times/day (total 400 mg/day) for 7 days. At this point, the study team will perform an interim analysis of the data. If our primary endpoint is not achieved we may revise our endpoints and/or if additional power is required, we may recruit up to an additional n=20 volunteers per group. This analysis may also serve as a stop-go checkpoint for continuation of the second phase of the study. If we do not see any effects of celecoxib on endothelial or cardiovascular function, we will not proceed to phase 2. If we do see a negative effect, we will proceed to phase 2.
  In phase 2 participants will be re-invited to the study site following a 4-8 week washout period. Participants will then receive either treatment with placebo + 10g L-arginine supplementation (20 participants) or celecoxib + 10g arginine supplementation (20 participants) for a total of 7 days
  Interventions: Drug: Celecoxib; Other: L-arginine + celecoxib
- Placebo (Placebo Comparator): Phase 1: Twenty volunteers will receive a placebo capsule, 2 times/day (total 400 mg/day) for 7 days. At this point, the study team will perform an interim analysis of the data. If our primary endpoint is not achieved we may revise our endpoints and/or if additional power is required, we may recruit up to an additional n=20 volunteers per group. This analysis may also serve as a stop-go checkpoint for continuation of the second phase of the study. If we do not see any effects of celecoxib on endothelial or cardiovascular function, we will not proceed to phase 2. If we do see a negative effect, we will proceed to phase 2.
  In phase 2 participants will be re-invited to the study site following a 4-8 week washout period. Participants will then receive either treatment with placebo + 10g L-arginine supplementation (20 participants) or celecoxib + 10g arginine supplementation (20 participants) for a total of 7 days
  Interventions: Other: Placebo; Other: L-arginine + placebo

INTERVENTIONS:
Drug: Celecoxib — Two 200 mg capsules per day (400 mg/day) for 7 days
  Other Names: Celebrex
  Arms: Celecoxib
Other: Placebo — 2 capsules/day for 7 days
  Arms: Placebo
Other: L-arginine + placebo — L-arginine = Five capsules of 2 mg per day (10 mg/day) for 7 days Placebo = 2 capsules/day for 7 days
  Arms: Placebo
Other: L-arginine + celecoxib — L-arginine = Five capsules of 2 mg per day (10 mg/day) Celecoxib = Two 200 mg capsules per day (400 mg/day) for 7 days
  Arms: Celecoxib

SUMMARY:
A single centre, placebo controlled, blinded (participant, investigator, outcome assessor) trial to evaluate the effects of COX-2 inhibition with celecoxib on endothelial function in healthy male volunteers.

DETAILED DESCRIPTION:
Primary Objective: To perform a systemic analysis of how COX-2 inhibition by celecoxib affects vascular function and 'omic biomarkers including those associated with the COX-2/prostacyclin/ADMA axis in healthy male volunteers

Secondary Objective: To investigate how this is altered by L-arginine supplementation

Methods: A single centre, double blind, placebo controlled trial will be carried out in healthy male volunteers between 18 and 40 years of age. In phase 1, participants will be blinded and randomised to receive either Celecoxib 200mgBD for 7 days or placebo. The primary endpoint is endothelial function measured by EndoPAT. In Phase 2, the same participants will receive either Celecoxib 200mgBD for 7 days + 10g L-arginine supplementation or placebo + 10g L-arginine supplementation to see if L-arginine can reverse any endothelial dysfunction caused by Celecoxib. Secondary outcomes will include measurement of 'omic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* No abnormal findings on medical history, screening physical examination, hematology, biochemistry, urinalysis (including specific gravity), and vital signs (sitting blood pressure, sitting pulse rate, sitting respiratory rate and body temperature) within 2 weeks of commencement of the study.
* Normal fasting lipid profile
* Non-smoking
* Clear venous access in upper limbs
* BMI: 18-30
* No history or signs of drug abuse
* No other medication 4 weeks before or during the study
* Informed written consent

Exclusion Criteria:

* Any history of allergy to NSAIDS or arginine
* Significant medical conditions
* Pulse rate <50 bpm
* Sitting systolic blood pressure <80 or >160 mmHg
* Sitting diastolic pressure <60 or >100 mmHg
* Baseline endothelial dysfunction (as defined by EndoPAT; LnRHI <0.51)
* Participation in other clinical study 8 weeks before or during the study
* Donation of blood 8 weeks before or during the study
* Those on medication that cannot be discontinued

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male Volunteers
Enrollment: 44 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Mitchell, Professor, Study Director — Imperial College London
Locations (1):
- Imperial College Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirkby NS, Zaiss AK, Urquhart P, Jiao J, Austin PJ, Al-Yamani M, Lundberg MH, MacKenzie LS, Warner TD, Nicolaou A, Herschman HR, Mitchell JA. LC-MS/MS confirms that COX-1 drives vascular prostacyclin whilst gene expression pattern reveals non-vascular sites of COX-2 expression. PLoS One. 2013 Jul 9;8(7):e69524. doi: 10.1371/journal.pone.0069524. Print 2013. PMID 23874970
- [Background] Kirkby NS, Chan MV, Zaiss AK, Garcia-Vaz E, Jiao J, Berglund LM, Verdu EF, Ahmetaj-Shala B, Wallace JL, Herschman HR, Gomez MF, Mitchell JA. Systematic study of constitutive cyclooxygenase-2 expression: Role of NF-kappaB and NFAT transcriptional pathways. Proc Natl Acad Sci U S A. 2016 Jan 12;113(2):434-9. doi: 10.1073/pnas.1517642113. Epub 2015 Dec 28. PMID 26712011
- [Background] Warner TD, Mitchell JA. COX-2 selectivity alone does not define the cardiovascular risks associated with non-steroidal anti-inflammatory drugs. Lancet. 2008 Jan 19;371(9608):270-3. doi: 10.1016/S0140-6736(08)60137-3. No abstract available. PMID 18207021
- [Background] Kirkby NS, Lundberg MH, Chan MV, Vojnovic I, Solomon AB, Emerson M, Mitchell JA, Warner TD. Blockade of the purinergic P2Y12 receptor greatly increases the platelet inhibitory actions of nitric oxide. Proc Natl Acad Sci U S A. 2013 Sep 24;110(39):15782-7. doi: 10.1073/pnas.1218880110. Epub 2013 Sep 3. PMID 24003163
- [Background] Ahmetaj-Shala B, Kirkby NS, Knowles R, Al'Yamani M, Mazi S, Wang Z, Tucker AT, Mackenzie L, Armstrong PC, Nusing RM, Tomlinson JA, Warner TD, Leiper J, Mitchell JA. Evidence that links loss of cyclooxygenase-2 with increased asymmetric dimethylarginine: novel explanation of cardiovascular side effects associated with anti-inflammatory drugs. Circulation. 2015 Feb 17;131(7):633-42. doi: 10.1161/CIRCULATIONAHA.114.011591. Epub 2014 Dec 9. PMID 25492024

RESULTS

PARTICIPANT FLOW:
Groups:
- Celecoxib: 22 participants were randomised and allocated to the celecoxib arm (200mg capsule taken orally twice a day for 7 days. Of these 2 participants withdrew from the study before the second study visit. In the final analysis there were 20 participants in the celecoxib arm.
- Placebo: 22 participants were randomised and allocated to the placebo arm (identical capsule to celecoxib containing placebo, 1 capsule taken orally twice daily for 7 days). Of these 2 participants were withdrawn from the study due to concomitant viral infection during the study week. In the final analysis there were 20 participants in the Placebo arm.
Period: Overall Study
Arm/Group | Celecoxib | Placebo
Started | 22 | 22
Completed | 20 | 20
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Celecoxib: Celecoxib
- Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (6) | 27.1 (6) | 26.8 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 20 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 10 | 20
  Asian | 4 | 7 | 11
  Oriental | 4 | 1 | 5
  Mixed | 1 | 0 | 1
  Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Log Reactive Hyperaemic Index
Description: Measured using the EndoPAT 2000 device (which is an FDA approved medical device).
  Data are issued by the equipment as:
  LnRHI (Log Reactive hyperaemic index), a reduction from the individual participant baseline value indicates endothelial dysfunction
Time Frame: Baseline and 7 days
Population: Data presented as mean change from baseline (delta)
Measure: Mean (Standard Deviation); unit: LnRHI (Log Reactive hyperaemic index)
Groups:
- Celecoxib: Celecoxib 200mg capsule taken orally twice a day for 7 days
- Placebo: Identical capsule to celecoxib containing placebo, 1 capsule taken orally twice daily for 7 days
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 20 | 20
LnRHI (Log Reactive hyperaemic index) | 0.003 (0.35) | 0.095 (0.33)

2. Primary Outcome: Augmentation Index
Description: Measured using the EndoPAT 2000 device (which is an FDA approved medical device) at baseline and at 7 days.
  Data are issued by the equipment. Augmentation index (which is a surrogate for vascular stiffness). An increase indicates an increase in vascular stiffness.
Time Frame: Baseline and 7 days
Measure: Mean (Standard Deviation); unit: Augmentation Index
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 20 | 20
Augmentation Index | 3.7 (9.05) | -2.54 (10.24)

3. Secondary Outcome: Blood Pressure
Description: Participants will record their blood pressure daily using a home monitoring device at rest on day 1 (baseline) and day 7. Reported as change in systolic blood pressure (delta) from baseline.
Time Frame: Baseline and 7 Days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 20 | 20
mmHg | -1.45 (11.8) | 2.03 (7.97)

4. Secondary Outcome: Increase/Decrease of Cardiovascular Biomarkers From Baseline
Description: Measured using mass spectrometry on serum samples collected at baseline and at 7 days.
Time Frame: Baseline and 7 days
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Celecoxib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT04765644/Prot_SAP_000.pdf